CLINICAL TRIAL: NCT05244109
Title: Bacterial Translocation in Spondyloarthritis: Evaluation Before and After Starting a Biomedicine.
Brief Title: Biomedicines and Bacterial Translocation in Spondyloarthritis
Acronym: TEARE-BIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021/577
Record Dates: First submitted 2022-01-27; First posted 2022-02-17 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-04

CONDITIONS: Axial Spondyloarthritis
Keywords: bacterial translocation
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NSAIDs (Experimental): Patients responding to any class of NSAIDs and unlikely to initiate biotherapy
  Interventions: Other: Blood sample
- Anti-TNF antibody (Experimental): Patients requiring the introduction of biotherapy according to current recommendations and randomized to the anti-TNF treatment arm
  Interventions: Other: Blood sample; Drug: anti-TNF antibody administration
- Anti-IL17 antibody (Experimental): Patients requiring the introduction of biotherapy according to current recommendations and randomized to the anti-IL-17 treatment arm
  Interventions: Other: Blood sample; Drug: anti-IL-17 antibody administration

INTERVENTIONS:
Other: Blood sample — Blood samples (2 times; 21mL per visit)
Drug: anti-TNF antibody administration — Anti-TNF antibody administration, according to current recommendations and randomization results
  Arms: Anti-TNF antibody
Drug: anti-IL-17 antibody administration — Anti-IL-17 antibody administration, according to current recommendations and randomization results
  Arms: Anti-IL17 antibody

SUMMARY:
The aim of this project is to evaluate the effect of anti-TNF and anti-IL17 biotherapies on bacterial translocation in patients with NSAID-resistant axial spondyloarthritis.

DETAILED DESCRIPTION:
Axial spondyloarthritis is a common inflammatory rheumatic disease and its management is based on the use of NSAIDs and biotherapies (anti-TNF and anti-IL17 antibodies). Its pathophysiology involves the digestive mucosa. The colon of patients with spondyloarthritis is the site of asymptomatic inflammation. This inflammation results from dysbiosis, which is responsible for activation of innate immunity linked to bacterial translocation phenomena. Dendritic cells are then activated and the immune response is polarized towards the IL23/Th17 axis. This translocation is secondary to an increase in colonic permeability. The increase in digestive permeability allows translocation of bacteria or bacterial fragments, primarily lipopolysaccharide (LPS).

Some proinflammatory cytokines (TNF, IFNγ, and IL23) cause an increase in digestive permeability. IL17 produced in the digestive mucosa has two different effects. Indeed, two types of colonic T cells produce IL17: regulatory T Helpers 17 producing IL10 and IL17 and inflammatory T Helpers 17 producing IL17 and IFNγ.

The investigators hypothesize that biotherapies decrease bacterial translocation. They suspect a lesser effect of anti-IL17 compared to anti-TNF because of the potential inhibition of Treg17 lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* Axial spondyloarthritis (2009 ASAS criteria)
* NSAID arm: Responding to any class of NSAID and not likely to initiate biotherapy
* anti-TNF/anti-IL-17 arms: Need to introduce a biomedical drug according to current recommendations (objective signs of inflammation, i.e. MRI sacroiliitis or increased CRP, and failure of two NSAIDs of different classes)

Exclusion Criteria:

* IBD already diagnosed by a gastroenterologist or suspicion of IBD (bloody diarrhea)
* Previous exposure to a biomedical drug (anti TNF or anti IL 17).
* Antibiotic use in the 3 months prior to inclusion
* Contraindications for treatment with anti-TNF or anti-IL17 (for all patients)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Difference in serum LPS concentration | 3 months
  Difference in serum LPS concentration, measured by liquid chromatography-mass spectrometry, between D0 (before anti-TNF or anti-IL 17) and D90

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No